CLINICAL TRIAL: NCT07196423
Title: Glutamate Changes as a New Neurocognitive Marker in Psychosis
Brief Title: Early Psychosis: Investigating Cognition
Acronym: EPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24048; 226715/Z/22/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2025-05-02; First posted 2025-09-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: First Episode Psychosis (FEP); Psychosis
Keywords: psychosis; cognition; glutamate; transcranial direct current stimulation; fMRS; first episode psychosis; GABA; working memory; magnetic resonance spectroscopy
MeSH Terms: conditions — Psychotic Disorders | interventions — Transcranial Direct Current Stimulation; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All participants in Study 1 will receive tDCS non-invasive brain stimulation. Participants in Study 2 will take part in an interview without any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study1a and 1b (Experimental): Study 1a: Will typically take place over 2-3 sessions (depending on participant's availability) spaced 1-7 days apart on average, and a 2-month follow up (FEP participants only). The first session (which could be split into two) will take approximately 4-5 hours in total consisting of several questionnaires, tasks, and up to 1 hour of MRI scanning. The second session will take approximately 2 hours and involve receiving tDCS stimulation and completing the cognitive task. The 2-month follow up will take up to 2 hours and involve assessing WM performance, symptoms scores (PANSS), CAPE-P15, quality of life and social and occupational functioning.
  Study 1b: Will take place on the same day as the second part of study 1a and will involve one additional scan of up to an hour in duration.
  Interventions: Device: Transcranial direct current stimulation (tDCS); Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — 2mA anodal stimulation to be delivered for 20 minutes using a Neuroconn DC stimulator PLUS which will be repeated once after a 20-minute break.
Diagnostic Test: Magnetic Resonance Imaging — Using a 7T Philips scanner with total scanning session lasting no more than 1 hour.

SUMMARY:
The project aims to explore changes in brain chemistry in individuals who have recently experienced psychosis. Recent research suggests that chemicals in the brain, specifically one called glutamate, may behave differently in people who have experienced psychosis compared to those who have not. It is also known that some individuals with psychosis can find tasks involving memory and attention more challenging. This study aims at understanding how brain chemistry is linked to memory and attention, and if this is different between people who have and have not experienced psychosis.

The study will also investigate how a commonly used brain stimulation technique might help people with psychosis and other conditions by altering brain chemistry for a very short period. Non-invasive brain stimulation using very weak electrical stimulation has been used to help improve symptoms in individuals with psychosis and many other conditions, and has been shown to alter brain chemistry for a few hours after stimulation. However, it does not work for everyone. It will be investigated if levels of glutamate can predict whether brain stimulation will help an individual or not. In other words, the study investigates if glutamate can be used as a marker for tailoring treatments.

This project also aims to collect personal experiences or challenges that individuals with psychosis face. This information will be gathered through interviews. This will help to understand what specific difficulties individuals have, such as with certain aspects of memory and attention. The interview will also gather opinions and concerns about brain imaging and brain stimulation and current understandings of chemicals in the brain. For example, the study will explore why individuals may not want to take part in brain imaging or brain stimulation.

DETAILED DESCRIPTION:
TRIAL / STUDY BACKGROUND INFORMATION AND RATIONALE

Cognitive impairment in psychosis:

Cognitive impairments occur in up to 80% of people living with psychosis. The recent landscape report, commissioned by the Wellcome Trust, highlighted that cognitive impairments are an "area of concern for people with psychosis" (p.36) and, furthermore, that "personalising the intervention approach...is desirable" (p.39). Specific cognitive symptoms are variable across individuals, but they are relevant for the individual as they predict day-to-day functioning and quality of life. Current interventions aiming at cognitive improvements are effective for some, but not all, individuals with psychosis. To increase the amount of viable and effective treatment options, a personalised approach based on improved understanding into the variability in cognitive impairments in psychosis is needed.

This project aims to explore perceptions of cognitive impairment & treatment from those with first-hand experience (Study 2); to explore a potential neurochemical marker (glutamate levels, in particular) for cognitive functioning with a focus on working memory (WM) (Study 1a); and to assess how this marker may predict changes in response to a single 'accelerated' session of non-invasive brain stimulation using transcranial direct current stimulation (tDCS) (Study 1a). Additionally, the study aims to explore the effects of accelerated tDCS on neurochemistry in individuals with first-episode psychosis (FEP; Study 1b). This 'accelerated' approach involves applying two stimulations in proximity during one testing session as recommended by several authors to safely maximise potential stimulation effects. The investigators chose tDCS as intervention method due to its potential for influencing glutamate levels (see below). Through these three interconnected studies using functional magnetic resonance spectroscopy (fMRS), transcranial direct current stimulation (tDCS) and interview approaches, the study aims at better understanding and informing potential future treatment options for cognitive impairment in psychosis.

It is important to note that while this study will use tDCS as part of this project, this is not an interventional study, in the respect that it is not assessing the impact of tDCS directly on symptoms or quality of life. In study 1a, the investigators will explore statistical relationships between changes in neurochemistry during the cognitive task, and changes in task performance during and following tDCS. In study 1b, the study will explore how neurochemistry is temporarily altered following accelerated tDCS in a subset of FEP participants. This will allow to validate previous work in healthy controls showing changes in Glu following tDCS, and to assess relationships between task performance and neurometabolite change. Thus, study 1a aims at establishing a link between neurochemical changes and subsequent responses to tDCS, while study 1b, aims to corroborate that tDCS has indeed influenced neurochemical changes in FEP individuals. Further details in the sections below.

Experience of cognitive impairment and perceptions of interventions in psychosis:

There is relatively little research exploring the subjective impact of cognitive impairments experienced through psychosis. Yet, impairments in cognitive functioning are experienced by 75-80% of people living with psychosis, and any future intervention that is designed to alleviate these impairments will have to target the most salient concerns of individuals with lived experiences to enhance uptake and engagement with the intervention. Past research that has interviewed individuals with psychosis has found impairments in cognitive functioning negatively impact on individuals daily functioning, including vocational performance, and on their self-concept, and relationships with others. Further interviews have shown that the notion of future interventions designed to enhance cognitive strengths has been received positively by individuals with psychosis. However, except for these studies little is known about this area, and these studies focused on young people (aged 18-26) receiving treatment in Australia. Additionally, relatively little is known about the perceptions of this demographic about views towards non-invasive brain stimulation approaches and use of magnetic resonance imaging in potential treatment plans. Study 2 will use semi-structured interviews to improve insights into the subjective impact of cognitive impairment and perceptions of non-invasive brain stimulation/ imaging among NHS patients in the UK. These will give valuable insights into what matters to patients and how potential interventions are perceived.

Working memory (WM) and psychosis:

Although several different cognitive functions can be affected in individuals with psychosis (perceptions of which will be explored in study 2), some cognitive domains seem particularly vulnerable, including associative processes in episodic and working memory (WM). WM is a crucial component of goal-directed behaviour. For instance, in a conversation we need to keep our semantic goals (the main message we want to convey) active in WM as well as a representation of what has been said already. Similarly, if we want to evaluate whether our actions have been successful and in line with our goals, i.e. monitoring our own performance, we need to keep a representation of the context and relevant information active in WM. These monitoring processes are often compromised in individuals with schizophrenia, thereby impacting goal-directed behaviour. Thus, impairments in WM are linked to impairments in goal-directed behaviour and will impact on a range of everyday life tasks.

Evidence from brain imaging studies using magnetic resonance spectroscopy (MRS) have given recent insights into the neurochemistry which underlies our ability to perform WM tasks and potential differences between those with and without psychosis. MRS is a specialised form of magnetic resonance imaging (MRI) which allows for quantification of neuro-metabolites, including glutamate (Glu) and GABA, which play a key role in regulating activity within the brain. Recent work has revealed a link between cognitive functions in schizophrenia and MRS measures of glutamate acquired at rest. In more dynamic measures taken during a cognitive task using fMRS, Jelen et al (2019) found that levels of Glu increase when transitioning from low to high WM conditions in healthy controls but not in individuals with psychosis. In Study 1a, we will build on the previous literature by using fMRS to explore how neurometabolites, including Glu, vary during a WM task between individuals with first episode psychosis and controls and how these modulations in task-dependent Glu-level modulations are related to the individual's WM performance.

Modulating glutamate using tDCS:

There is some evidence that Glu levels in the brain may be related to treatment outcome. A recent meta-analysis showed increased medial frontal Glu levels in treatment-resistant psychosis but decreased Glu levels in treatment responders, indicating a preliminary association between Glu levels and treatment outcome. Therefore, it seems to be promising to further investigate the relationship between Glu levels, cognitive functions, and treatment outcomes.

After establishing how Glu changes in response to a WM task in both first episode psychosis (FEP) individuals and health controls, the study aims to evaluate if this natural flexibility in Glu is related to changes in Glu driven by external means which could be developed into robust therapies in the future. Specifically, Study 1a will explore the potential relationship between Glu change during the WM task and behavioural change attributed to transcranial direct current stimulation (tDCS). The investigators will then extend this in Study 1b to corroborate if Glu levels have indeed been modulated by exposure to tDCS.

Transcranial direct-current stimulation (tDCS) is a non-invasive brain stimulation method which can modulate Glu levels in stimulated brain areas. A weak current is applied to the scalp influencing the underlying cortex by altering the membrane potential of neurons proximal to the surface electrode. Anodal stimulation is frequently reported to increase the cortical excitability which can induce increased neural plasticity and thereby lead to functional changes that last longer than the actual stimulation. TDCS has the advantage that it can modulate Glu levels in targeted brain areas and, compared to many pharmacological interventions, has relatively mild and short-lasting side effects (e.g. tingling sensations), has demonstrated good tolerability within the majority of patient groups and has the potential to develop for home use in the future.

TDCS has already been used in individuals with schizophrenia to improve executive functions and learning as well as working memory and clinical symptoms. Although the effect sizes of tDCS stimulations are often noted to be variable within healthy individuals, studies in several different brain regions have shown links between relevant task performance and tDCS response.

The investigators propose that task-related Glu changes (measured with fMRS) predict more precisely who will benefit most from tDCS stimulation. The investigators will assess this in Study 1a through evaluating the relationship between fMRS measured Glu change during a WM task and performance change in the same take following tDCS. In a subset of participants (Study 1b), the study will additionally explore any change in fMRS measured Glu immediately following tDCS. Thus, the study will investigate the relationship between pre- and post-tDCS Glu modulations, within-task Glu modulations and behavioural task performance.

The aim in Study 1b is not to evaluate the effectiveness of tDCS (this would need to be tested in a follow-up RCT), but to establish the relationship between Glu dynamics in a cognitive task and the effect of an intervention that modulates the Glu system. The study involves a CE marked device which has been used extensively for research purposes.

The investigators do not anticipate that any of our results will affect future clinical practice directly, however, the information gathered form the various sub-studies will provide valuable knowledge that could provide the foundation for future intervention developments.

ELIGIBILITY:
Inclusion Criteria for FEP Group (studies 1a and 1b):

Eligibility criteria for first episode psychosis group are as follows:

1. Aged 18-55 years.
2. Ability to understand and willing to give written informed consent.
3. Fluent in English to be able to understand all cognitive task instructions and questionnaires.
4. Current psychotic disorder of less than 5yrs total duration. Defined as meeting DSM-5 criteria consistent with a diagnosis of schizophrenia, schizoaffective disorder, bipolar affective disorder, or severe depression with psychosis.
5. At least 8 weeks of stable treatment.
6. Ability to travel to the University of Nottingham for in-person testing.

Exclusion Criteria for FEP Group (Studies 1a and 1b):

1. Clinically significant neurological or comorbid psychiatric disorder in the opinion of the investigator.
2. History of clinically significant head injury
3. Current harmful use of, or dependence on, psychoactive substances (excluding nicotine) in the opinion of the investigator
4. Current use of any medication which may interfere with the study in the opinion of the investigator, i.e. any medication that might affect the neurochemicals of interest
5. Contraindications for MR scanning as assessed by SPMIC screening form and trained scanner operator (e.g. claustrophobia, pregnancy, metal implants, etc.)
6. Contraindications for transcranial direct current stimulation as assessed by standard screening form (e.g. cardiac pacemaker or other implanted devices, seizures, epilepsy, open head wound, etc.)
7. Having taken part within the previous month as a participant in a clinical trial that involved taking a drug or having an invasive procedure.

Inclusion Criteria for Healthy Matched Controls (Studies 1a and 1b):

Matched healthy control participants will be recruited from a local database of volunteers, from posters and online advertisements.

Inclusion criteria (matched controls):

1. Aged 18 - 55 years.
2. Ability to understand and willing to give written informed consent.
3. English as first language or fluent in English.
4. Ability to travel to the University of Nottingham for in-person testing.

Exclusion criteria for Health Matched Controls (Studies 1a and 1b):

1. Personal or family history of psychosis.
2. Clinically significant neurological or psychiatric disorder.
3. History of clinically significant head injury.
4. Current harmful use of, or dependence on, psychoactive substances (excluding nicotine and caffeine) in the opinion of the investigator.
5. Current use of any medication, which may interfere with the study in the opinion of the investigator i.e. any medication that might affect the neurochemicals of interest.
6. Contraindications for MR scanning as assessed by SPMIC screening form and trained scanner operator (e.g. claustrophobia, pregnancy etc).
7. Contraindications for transcranial direct current stimulation as assessed by standard screening form (e.g. cardiac pacemaker or other implanted devices, seizures, epilepsy, open head wound, etc.)
8. Having taken part within the previous month as a participant in a clinical trial that involved taking a drug, being paid an inconvenience allowance, or having an invasive procedure (e.g. venepuncture >50ml, endoscopy).

Inclusion Criteria for participants with lived experiences of psychosis (Study 2):

1. Aged 18+ years.
2. Ability to understand and willing to give written informed consent.
3. Fluent in English to be able to understand and answer all questions.
4. History of psychotic disorder defined as DSM-5 criteria for diagnosis of schizophrenia, schizoaffective disorder, bipolar affective disorder, or severe depression with psychosis. No limit of time since first episode.
5. At least 8 weeks of stable treatment.
6. Ability to travel to the University of Nottingham for in-person testing.

Exclusion Criteria for participants with lived experiences of psychosis (Study 2):

1. Clinically significant neurological or comorbid psychiatric disorder.
2. Current harmful use of, or dependence on, psychoactive substances (excluding nicotine) in the opinion of the investigator.
3. Having taken part within the previous month as a participant in a clinical trial that involved taking a drug or having an invasive procedure.
4. Lived experience where psychosis symptoms have not been directly experienced by the individual (e.g., support or carer role to someone else).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Measures of glutamate and GABA change (quantified using fMRS) during a working memory task | Day 1, during fMRS scan, blocks with working memory task vs. blocks with control task.
  Difference in glutamate and GABA levels between different phases/WM load in a working memory task (Study 1a).
Correlation between glutamate and GABA responses during a WM task and tDCS outcome (accuracy) | within 1 week
  Neurometabolite changes during a WM task (as described above, outcome measure 1) will be correlated with changes in accuracy in a WM task after tDCS brain stimulation.
Correlation between glutamate and GABA responses during a WM task and tDCS outcome (reaction time) | within 1 week
  Neurometabolite changes during a WM task (as described above, outcome measure 1) will be correlated with changes in reaction times in a WM task after tDCS brain stimulation.
Qualitative data analysis: Perceived cognitive impairments in psychosis | Study day 2
  Thematic analysis of impact of experiencing cognitive impairments (or perceived improvements) on individuals' lives in semi-structured interviews (Study 2).
Qualitative data analysis: Expectations and concerns around interventions that involve brain scanning and brain stimulation | Study day 2
  Themes (as outcome of a thematic analysis) that describe FEP participants' interests and expectations for future interventions designed to alleviate the impact of cognitive impairments, particularly regarding any future interventions using non-invasive brain stimulation methods (Study 2). Data will be collected in a semi-structured interview.

SECONDARY OUTCOMES:
Difference in glutamate levels during working memory task pre- and post-tDCS stimulation | within 1 week (pre- and post-tDCS fMRS acquisitions; post-tDCS scan will take place immediately after tDCS stimulation)
  Glutamate concentration in the medial frontal cortex while the participant is engaged in an associative working memory task pre-tDCS stimulation vs. post-tDCS stimulation
Difference in GABA levels during working memory task pre- and post-tDCS stimulation | within 1 week (pre- and post-tDCS fMRS acquisitions; post-tDCS scan will take place immediately after tDCS stimulation)
  GABA concentration in the medial frontal cortex while the participant is engaged in an associative working memory task pre-tDCS stimulation vs. post-tDCS stimulation
Changes in other neurometabolites (tCR, GSH) during different phases of a working memory task. | Day 1, during fMRS scan, blocks with working memory task vs. blocks with control task.
  Level of neurometabolite concentration (tCR, GSH) in the medial frontal cortex during the associative Working Memeory task as compared to a control condition without working memory load in individuals with psychosis and matched controls.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and psychosis symptom severity (PANSS). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with symptom scores from PANSS.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and psychosis symptom severity (SPS). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with symptom scores from Scale of Prodromal Symptoms (SPS).
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and psychosis symptom severity (CAPE-P15). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with symptom scores from the Community Assessment of Psychic Experiences (CAPE-P15).
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and socio-occupational performance (PSP). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with scores from the Personal and Social Performance Scale (PSP).
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and quality of life (WHOQOL-BREF). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with quality of life scores from the World Health Organisation Quality of Life Brief Version (WHOQOL-BREF).
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and experience of disability (WHODAS 2.0) | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with disability assessment scores from the World Health Organisation Disability Assessment Schedule (WHODAS 2.0).
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task and autism spectrum symptoms (AQ-50). | Within 2 months from first fMRS acquisition
  Neurometabolite concentration changes during an associative WM task will be correlated with scores from the Autism Quotient - 50 item questionnaire.
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and accuracy in a change detection working memory task. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with accuracy (percentage of correct answers) in a change detection working memory task.
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and performance in the forward/backward number span task. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with the individual's number span (maximum number of numbers correctly recalled).
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and performance in the Corsi block test. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with the individual's block span (maximum number of blocks correctly recalled).
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and processing speed. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with processing speed as measured in the digit-symbol substitution test (number of correctly associated items in a fixed amount of time).
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and processing speed (simple and choice reaction time). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with processing speed as measured with a simple and a choice reaction time (RT) task (RT in simple RT task, difference in RT between choice RT task and simple RT task).
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and processing speed/attentional shifting (Trail Making Test). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with processing speed/attentional shifting performance as measured with the Trail Making Test (TMT, completion time).
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and cognitive control (interference). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with interference reaction times (difference between incongruent and congruent trial reaction times) in a cognitive control task.
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and performance monitoring. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with the error rate in a cognitive control task.
Correlation of neurometabolite concentration levels (glutamate, GABA) during rest (static MRS) and meta-cognitive monitoring. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration levels at rest (static MRS) will be correlated with the percentage of perceived errors (relative to unperceived errors) in an error awareness task.
Correlation between WM performance and visual imagery scores (VVIQ) | WM performance and VVIQ will be acquired within 10 days.
  Correlation between accuracy in the associative visual WM task and visual imagery scores as measured with the Vividness of Visual Imagery Questionnaire (VVIQ).
Correlation between WM performance and visual imagery scores (SUIS) | WM performance and SUIS will be acquired within 10 days.
  Correlation between accuracy in the associative visual WM task and visual imagery scores as measured with the Spontaneous Use of Imagery Scale (SUIS).

OTHER OUTCOMES:
Alignment between objective cognitive measures and subjective experiences of cognitive impairments | Study day 2
  Qualitative data analysis: the self-reported cognitive strengths and deficits in Study 2 will be compared to the cognitive performance profile (accuracy, RTs, completion times) in working memory, attentional and cognitive control tasks from Study 1. This will be done on an individual case basis.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task (fMRS) and accuracy in a change detection working memory task. | Within 2 months of MRS data acquisition.
  Neurometabolite concentration during the associative working memory task (fMRS, percent change in neurometabolite level between WM task and control condition) will be correlated with accuracy (percentage of correct answers) in a change detection working memory task.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task (fMRS) and processing speed (digit-symbol substitution task). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration during the associative working memory task (fMRS, percent change in neurometabolite level between WM task and control condition) will be correlated with number of correctly associated items in the digit-symbol substitution task.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task (fMRS) and processing speed (simple and choice RT). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration during the associative working memory task (fMRS, percent change in neurometabolite level between WM task and control condition) will be correlated with reaction times in a simple RT task and the difference in reaction times between a simple and a choice RT task.
Correlation of neurometabolite concentration changes (glutamate, GABA) during WM task (fMRS) and processing speed/attentional shifting (Trail Making Test). | Within 2 months of MRS data acquisition.
  Neurometabolite concentration during the associative working memory task (fMRS, percent change in neurometabolite level between WM task and control condition) will be correlated with the completion times in the Trail Making Test.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Danielmeier, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Magnetic resonance spectroscopy (MRS/fMRS) data functional MRI data Performance on cognitive assessments at different study time points QoL and other questionnaire data interview transcripts or summarised interview data (depending on participant consent)
Time Frame: Data will be shared after publication of the study results. Data shared in OSF and UK Data Service do not have a time limitation.
Access Criteria: IPD from study 1a and b will be uploaded to OSF. Interview data will be deposited with the UK data service.

REFERENCES:
- [Background] Russo R, Wallace D, Fitzgerald PB, Cooper NR. Perception of comfort during active and sham transcranial direct current stimulation: a double blind study. Brain Stimul. 2013 Nov;6(6):946-51. doi: 10.1016/j.brs.2013.05.009. Epub 2013 Jun 25. PMID 23835166
- [Background] Hill AT, Fitzgerald PB, Hoy KE. Effects of Anodal Transcranial Direct Current Stimulation on Working Memory: A Systematic Review and Meta-Analysis of Findings From Healthy and Neuropsychiatric Populations. Brain Stimul. 2016 Mar-Apr;9(2):197-208. doi: 10.1016/j.brs.2015.10.006. Epub 2015 Oct 23. PMID 26597929
- [Background] Yamada Y, Sumiyoshi T. Neurobiological Mechanisms of Transcranial Direct Current Stimulation for Psychiatric Disorders; Neurophysiological, Chemical, and Anatomical Considerations. Front Hum Neurosci. 2021 Feb 4;15:631838. doi: 10.3389/fnhum.2021.631838. eCollection 2021. PMID 33613218
- [Background] Morey-Nase C, Phillips LJ, Bryce S, Hetrick S, Wright AL, Caruana E, Allott K. Subjective experiences of neurocognitive functioning in young people with major depression. BMC Psychiatry. 2019 Jul 4;19(1):209. doi: 10.1186/s12888-019-2197-1. PMID 31272419
- [Background] Reinhart RM, Zhu J, Park S, Woodman GF. Medial-Frontal Stimulation Enhances Learning in Schizophrenia by Restoring Prediction Error Signaling. J Neurosci. 2015 Sep 2;35(35):12232-40. doi: 10.1523/JNEUROSCI.1717-15.2015. PMID 26338333
- [Background] Reinhart RM, Zhu J, Park S, Woodman GF. Synchronizing theta oscillations with direct-current stimulation strengthens adaptive control in the human brain. Proc Natl Acad Sci U S A. 2015 Jul 28;112(30):9448-53. doi: 10.1073/pnas.1504196112. Epub 2015 Jun 29. PMID 26124116
- [Background] Pilloni G, Charvet LE, Bikson M, Palekar N, Kim MJ. Potential of Transcranial Direct Current Stimulation in Alzheimer's Disease: Optimizing Trials Toward Clinical Use. J Clin Neurol. 2022 Jul;18(4):391-400. doi: 10.3988/jcn.2022.18.4.391. PMID 35796264
- [Background] Pena-Gomez C, Sala-Lonch R, Junque C, Clemente IC, Vidal D, Bargallo N, Falcon C, Valls-Sole J, Pascual-Leone A, Bartres-Faz D. Modulation of large-scale brain networks by transcranial direct current stimulation evidenced by resting-state functional MRI. Brain Stimul. 2012 Jul;5(3):252-263. doi: 10.1016/j.brs.2011.08.006. Epub 2011 Sep 5. PMID 21962981
- [Background] Moran EK, Gold JM, Carter CS, MacDonald AW 3rd, Ragland JD, Silverstein SM, Luck SJ, Barch DM. Both unmedicated and medicated individuals with schizophrenia show impairments across a wide array of cognitive and reinforcement learning tasks. Psychol Med. 2022 Apr;52(6):1115-1125. doi: 10.1017/S003329172000286X. Epub 2020 Aug 17. PMID 32799938
- [Background] Mondino M, Poulet E, Brunelin J. Moving to accelerated protocols of tDCS in schizophrenia: A case report. Brain Stimul. 2021 Jul-Aug;14(4):822-824. doi: 10.1016/j.brs.2021.05.006. Epub 2021 May 19. No abstract available. PMID 34022429
- [Background] Koolschijn RS, Emir UE, Pantelides AC, Nili H, Behrens TEJ, Barron HC. The Hippocampus and Neocortical Inhibitory Engrams Protect against Memory Interference. Neuron. 2019 Feb 6;101(3):528-541.e6. doi: 10.1016/j.neuron.2018.11.042. Epub 2018 Dec 20. PMID 30581011
- [Background] Hunter MA, Coffman BA, Gasparovic C, Calhoun VD, Trumbo MC, Clark VP. Baseline effects of transcranial direct current stimulation on glutamatergic neurotransmission and large-scale network connectivity. Brain Res. 2015 Jan 12;1594:92-107. doi: 10.1016/j.brainres.2014.09.066. Epub 2014 Oct 12. PMID 25312829
- [Background] Heimrath K, Brechmann A, Blobel-Luer R, Stadler J, Budinger E, Zaehle T. Transcranial direct current stimulation (tDCS) over the auditory cortex modulates GABA and glutamate: a 7 T MR-spectroscopy study. Sci Rep. 2020 Nov 18;10(1):20111. doi: 10.1038/s41598-020-77111-0. PMID 33208867
- [Background] Bystad M, Storo B, Gundersen N, Wiik IL, Nordvang L, Gronli O, Rasmussen ID, Aslaksen PM. Can accelerated transcranial direct current stimulation improve memory functions? An experimental, placebo-controlled study. Heliyon. 2020 Oct 3;6(10):e05132. doi: 10.1016/j.heliyon.2020.e05132. eCollection 2020 Oct. PMID 33033765
- [Result] Valiengo LDCL, Goerigk S, Gordon PC, Padberg F, Serpa MH, Koebe S, Santos LAD, Lovera RAM, Carvalho JB, van de Bilt M, Lacerda ALT, Elkis H, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation for Treating Negative Symptoms in Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):121-129. doi: 10.1001/jamapsychiatry.2019.3199. PMID 31617873
- [Result] Ullsperger M, Danielmeier C, Jocham G. Neurophysiology of performance monitoring and adaptive behavior. Physiol Rev. 2014 Jan;94(1):35-79. doi: 10.1152/physrev.00041.2012. PMID 24382883
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Orlov ND, Tracy DK, Joyce D, Patel S, Rodzinka-Pasko J, Dolan H, Hodsoll J, Collier T, Rothwell J, Shergill SS. Stimulating cognition in schizophrenia: A controlled pilot study of the effects of prefrontal transcranial direct current stimulation upon memory and learning. Brain Stimul. 2017 May-Jun;10(3):560-566. doi: 10.1016/j.brs.2016.12.013. Epub 2016 Dec 28. PMID 28057452
- [Result] Nakahara T, Tsugawa S, Noda Y, Ueno F, Honda S, Kinjo M, Segawa H, Hondo N, Mori Y, Watanabe H, Nakahara K, Yoshida K, Wada M, Tarumi R, Iwata Y, Plitman E, Moriguchi S, de la Fuente-Sandoval C, Uchida H, Mimura M, Graff-Guerrero A, Nakajima S. Glutamatergic and GABAergic metabolite levels in schizophrenia-spectrum disorders: a meta-analysis of 1H-magnetic resonance spectroscopy studies. Mol Psychiatry. 2022 Jan;27(1):744-757. doi: 10.1038/s41380-021-01297-6. Epub 2021 Sep 28. PMID 34584230
- [Result] Kirschner H, Klein TA. Beyond a blunted ERN - Biobehavioral correlates of performance monitoring in schizophrenia. Neurosci Biobehav Rev. 2022 Feb;133:104504. doi: 10.1016/j.neubiorev.2021.12.027. Epub 2021 Dec 16. PMID 34922988
- [Result] Katz B, Au J, Buschkuehl M, Abagis T, Zabel C, Jaeggi SM, Jonides J. Individual Differences and Long-term Consequences of tDCS-augmented Cognitive Training. J Cogn Neurosci. 2017 Sep;29(9):1498-1508. doi: 10.1162/jocn_a_01115. Epub 2017 Mar 2. PMID 28253083
- [Result] Habtewold TD, Rodijk LH, Liemburg EJ, Sidorenkov G, Boezen HM, Bruggeman R, Alizadeh BZ. A systematic review and narrative synthesis of data-driven studies in schizophrenia symptoms and cognitive deficits. Transl Psychiatry. 2020 Jul 21;10(1):244. doi: 10.1038/s41398-020-00919-x. PMID 32694510
- [Result] Gold JM. Cognitive deficits as treatment targets in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):21-8. doi: 10.1016/j.schres.2004.09.008. PMID 15531404
- [Result] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Result] Au, J., Karsten, C., Buschkuehl, M., &amp;amp;amp;amp; Jaeggi, S. M. (2017). Optimizing transcranial direct current stimulation protocols to promote long-term learning. Journal of Cognitive Enhancement, 1(1), 65-72.
- [Result] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Result] Wright, A. L., Phillips, L. J., Bryce, S., Morey-Nase, C., & Allott, K. (2019). Subjective experiences of cognitive functioning in early psychosis: a qualitative study. Psychosis, 11(1), 63-74.
- See also: Study website — https://the-epic-study.quarto.pub/the-epic-project/